CLINICAL TRIAL: NCT01344031
Title: A Phase 1 Trial of MK-2206 in Combination With Anastrozole, Fulvestrant, or Anastrozole Plus Fulvestrant in Postmenopausal Women With Estrogen Receptor Positive Metastatic Breast Cancer
Brief Title: MK2206 in Combination With Anastrozole, Fulvestrant, or Anastrozole and Fulvestrant in Treating Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02586; NCI-2011-02586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 201010701; WU-201010701; CDR0000699394; 201010701 (Other: Washington University School of Medicine); 8762 (Other: CTEP); N01CM00099 (NIH); P30CA091842 (NIH)
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-05

CONDITIONS: Estrogen Receptor Positive; Invasive Breast Carcinoma; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — MK 2206; Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (anastrozole and Akt inhibitor MK2206) (Experimental): Patients receive anastrozole PO on days 1-28. Beginning in course 2, patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: As of 8/19/2015, patients no longer receive Akt inhibitor MK2206.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Anastrozole; Other: Laboratory Biomarker Analysis
- Arm B (Akt inhibitor MK2206 and anastrozole) (Experimental): The RPTD of Akt inhibitor MK2206 with anastrozole is determined after 3 courses, administered as in Arm A.
  NOTE: As of 8/19/2015, patients no longer receive Akt inhibitor MK2206.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Anastrozole; Other: Laboratory Biomarker Analysis
- Arm C (Akt inhibitor MK2206 and fulvestrant) (Experimental): Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22, fulvestrant IM on day 1and day 15 of course 1 and then on day 1 of each course in each subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: As of 8/19/2015, patients no longer receive Akt inhibitor MK2206.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis
- Arm D (Akt inhibitor MK2206, anastrozole, fulvestrant) (Experimental): Patients receive Akt inhibitor MK2206 PO as in Arm A, anastrozole PO on days 1-28 and fulvestrant IM on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: As of 8/19/2015, patients no longer receive Akt inhibitor MK2206.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Anastrozole; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
  Arms: Arm A (anastrozole and Akt inhibitor MK2206); Arm B (Akt inhibitor MK2206 and anastrozole); Arm D (Akt inhibitor MK2206, anastrozole, fulvestrant)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
  Arms: Arm C (Akt inhibitor MK2206 and fulvestrant); Arm D (Akt inhibitor MK2206, anastrozole, fulvestrant)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of MK 2206 (Akt inhibitor MK2206) when given with anastrozole, fulvestrant, or anastrozole and fulvestrant in treating postmenopausal women with breast cancer that has spread to other parts of the body. Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole or fulvestrant may fight breast cancer by lowering the amount of estrogen the body makes. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving Akt inhibitor MK2206 together with anastrozole, fulvestrant, or anastrozole and fulvestrant may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of MK-2206 in combination with anastrozole based on toxicities observed during cycle 1 therapy. (Phase IA) II. To evaluate the tolerability of prolonged administration (3 months) of MK-2206 in combination with anastrozole at the MTD defined in Phase IA. (Phase IB) III. To determine the recommended phase II treatment dosing (RPTD) of MK-2206 in combination with anastrozole based on toxicities observed with prolonged drug administration. (Phase IB) IV. To determine the tolerability of fulvestrant (Arm C), or fulvestrant plus anastrozole (Arm D), respectively, in combination with MK-2206 (at the RPTD defined in Phase 1B). (Arms C and D) V. To determine the recommended phase II treatment dose (RPTD) of fulvestrant (Arm C) or fulvestrant plus anastrozole (Arm D), respectively, in combination with MK-2206 based on toxicities observed with prolonged drug administration (3 months). (Arms C and D) VI. To evaluate the toxicity profile of MK-2206 in combination with fulvestrant (Arm C) or fulvestrant plus anastrozole (Arm D), respectively, with prolonged drug administration. (Arms C and D)

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of MK-2206 in combination with anastrozole, or fulvestrant, or anastrozole plus fulvestrant.

II. To evaluate the clinical benefit rate (CBR: complete response [CR]+partial response [PR]+stable disease [SD] > 6 months), response rate (CR+PR), and percent of patients progression free at 6 months with the treatment of MK-2206 in combination with anastrozole, or fulvestrant or anastrozole plus fulvestrant in patients with estrogen receptor positive (ER+) metastatic breast cancer.

III. To examine serum levels of estradiol prior to and following 1 cycle of MK-2206 therapy.

TERTIARY OBJECTIVES:

I. To examine baseline tumor specimens for alterations in phosphatidylinositol 3 kinase (PI3K) and other pathway genes and to explore their relationship with treatment response.

II. To evaluate the effect of MK-2206 on tumor cell v-akt murine thymoma viral oncogene homolog 1 (AKT) signaling, proliferation, and apoptosis using serially collected tumor samples in available cases.

III. To examine changes in tumor cell glucose uptake by positron emission tomography (PET) with 2-[18F]fluoro-2-deoxy-D-glucose (FDG) at baseline and 24 h post day 1 MK-2206. (Phase IA) IV. To examine the phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutation status in circulating deoxyribonucleic acid (DNA) at baseline and following study therapy and to correlate with tumor tissue PIK3CA status and treatment response.

OUTLINE: This is a phase I, dose-escalation study of Akt inhibitor MK2206 followed by a recommended phase II dose (RPTD) study. Patients are assigned to the treatment arm that is currently open.

ARM A: Patients receive anastrozole orally (PO) on days 1-28. Beginning in course 2, patients receive Akt inhibitor MK-2206 PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: The RPTD of Akt inhibitor MK2206 with anastrozole is determined after 3 courses, administered as in Arm A.

ARM C: Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22, fulvestrant intramuscularly (IM) on day 1 and day 15 of course 1 and then on day 1 of each course in each subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive Akt inhibitor MK2206 PO as in Arm A, anastrozole PO on days 1-28 and fulvestrant IM on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: As of 8/19/2015, in all Arms, patients no longer receive Akt inhibitor MK2206.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer that is metastatic stage IV or recurrent metastatic (histologic/cytologic confirmation of recurrence preferred, but not required)
* Either the primary or the metastatic tumor must be positive for estrogen-receptor (> 1% tumor cell staining by immunohistochemistry or an Allred score of >= 3 by immunohistochemistry)
* Patient must have measurable or non-measurable lesions (defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria)

  * Note: to be eligible for the FDG PET imaging studies in Phase IA, the presence of measurable lesions of at least 1.5 cm or the presence of bone lesions is required
* Patients may have undergone any number of prior lines of chemotherapy or endocrine regimens but must not have a history of disease progression on anastrozole (Phase IA and Phase IB), fulvestrant (Arm C), or both anastrozole and fulvestrant (Arm D)

  * Phase IA and IB:

    * Currently being treated with anastrozole with no evidence of disease progression OR
    * Currently being treated with letrozole or exemestane with no evidence of disease progression and willing to switch to anastrozole for study enrollment OR
    * Considering switching to anastrozole due to disease progression from the most recent anti-cancer therapy
  * Arm C:

    * Currently being treated with fulvestrant with no evidence of disease progression OR
    * Considering switching to fulvestrant due to disease progression from the most recent anti-cancer therapy
  * Arm D:

    * Currently being treated with either anastrozole or fulvestrant with no evidence of disease progression OR
    * Currently being treated with letrozole or exemestane with no evidence of disease progression and willing to switch to anastrozole for study enrollment
    * Considering switching to anastrozole or fulvestrant due to disease progression from the most recent anti-cancer therapy
* Patients must be postmenopausal women as defined by one of the following:

  * Women > 60 years
  * Women =< 60 years with spontaneous cessation of menses > 12 months prior to registration
  * Women =< 60 years with cessation of menses of duration < 12 months or secondary to hysterectomy AND an follicle stimulating hormone (FSH) level in the postmenopausal range according to institutional standards (or > 34.4 IU/L if institutional range is not available) prior to registration
  * Women =< 60 years on hormonal replacement therapy who have discontinued hormonal therapy AND an FSH level in the postmenopausal range according to institutional standards (or > 34.4 IU/L if institutional range is not available) prior to registration
  * Status post bilateral surgical oophorectomy
  * Premenopausal women on a gonadotropin-releasing hormone (GnRH) analog
* Patients must have a life expectancy greater than 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin not above the institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine not above the institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* If patients have diabetes mellitus, fasting glucose must be =< 120 mg/dL and hemoglobin (Hb)A1c =< 8%
* Women of childbearing potential must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, the patient should inform the treating physician immediately
* Patients with known brain metastases are eligible if stable (no evidence of local progression) >= 3 months after local therapy and are off steroid
* Patients who are eligible for this study may also be eligible for and participate in National Cancer Institute (NCI) Protocol 9167, titled "Positron Emission Tomography (PET) with 18F-Fluoroestradiol (FES) as a Predictor of Response in Patients with Breast Cancer Scheduled to Be Treated with MK-2206 in Combination with Either an Aromatase Inhibitor or Fulvestrant on NCI Protocol 8762," in which case the FES-PET in Protocol 9167 has to be performed a minimum of 48 hours and a maximum of 30 days before the first dose of MK-2206; in addition, all FES-related side effects must have resolved before the first dose of MK-2206
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study; patient must have recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients may not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in the study
* Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP 450 3A4) are ineligible

  * Note: one week washout period is required in patients who were previously taking strong inhibitors or inducers of CYP450 3A4; patients who are currently taking moderate inhibitors or inducers of CYP450 3A4 are encouraged to switch to other medications that do not interact with CYP450 3A4
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial (i.e. HbA1c =< 8% and fasting glucose =< 120 mg/dL)
* Cardiovascular: baseline QT Fridericia formula (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Patients may not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing patients are excluded from the study
* Patients with known human immunodeficiency virus (HIV) positive status are excluded from this study
* Patients may not have had disease progression on anastrozole (Phase IA and Phase IB), fulvestrant (Arm C), both anastrozole and fulvestrant (Arm D) in either the neoadjuvant, adjuvant (defined as disease recurrence identified within 6 months of adjuvant discontinuation), or metastatic setting
* Patients may not have had grade 3 or intolerable grade 2 adverse events during run-in aromatase inhibitor (AI) or fulvestrant therapy prior to starting MK-2206
* Patients may not have had prior therapy with an AKT inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04-21 (Actual); Primary Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
MTD of Akt inhibitor MK-2206 in combination with anastrozole determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) (Phase IA) | 4 weeks
  Data analysis for the study will be descriptive in nature. Demographic and clinical characteristics of the subjects, toxicity by grade, adverse events, serious adverse events and death will be listed and summarized using descriptive statistics for each dose level.
RPTD of Akt inhibitor MK-2206 in combination with anastrozole evaluated by the tolerability of prolonged administration at the MTD assessed by CTCAE v4.0 (Phase IB) | 3 months
  Data analysis for the study will be descriptive in nature. Demographic and clinical characteristics of the subjects, toxicity by grade, adverse events, serious adverse events and death will be listed and summarized using descriptive statistics for each dose level.
RPTD of fulvestrant in combination with Akt inhibitor MK-2206 assessed by CTCAE v4.0 (ARM C) | 3 months
  Data analysis for the study will be descriptive in nature. Demographic and clinical characteristics of the subjects, toxicity by grade, adverse events, serious adverse events and death will be listed and summarized using descriptive statistics for each dose level.
RPTD of anastrozole plus fulvestrant in combination with Akt inhibitor MK-2206 assessed by CTCAE v4.0 (ARM D) | 3 months
  Data analysis for the study will be descriptive in nature. Demographic and clinical characteristics of the subjects, toxicity by grade, adverse events, serious adverse events and death will be listed and summarized using descriptive statistics for each dose level.

SECONDARY OUTCOMES:
Incidence of toxicity, assessed by CTCAE v4.0 | Up to 30 days post-treatment
Clinical benefit rate (CR+PR+SD for more than 6 months) | Up to 30 days post-treatment
Serum levels of estradiol prior to and following 1 course of Akt inhibitor MK-2206 therapy | Up to day 28

OTHER OUTCOMES:
Change in PI3K pathway abnormalities | Baseline up to 30 days post-treatment
Tumor cell AKT signaling | Up to 30 days post-treatment
  Descriptive statistics will be calculated for each dose level.
Tumor cell proliferation | Up to 30 days post-treatment
  Descriptive statistics will be calculated for each dose level.
Tumor cell apoptosis | Up to 30 days post-treatment
  Descriptive statistics will be calculated for each dose level.
Changes in tumor cell glucose uptake by 2-[18F]fluoro-2-deoxy-D-glucose (FDG)/PET | Baseline up to 24 hours post day 1 Akt inhibitor MK2206
  Descriptive statistics will be calculated for each dose level. The associations between changes in standardized uptake value (SUV) and clinical outcomes will also be explored graphically.
Change in PIK3CA mutation status in circulating DNA | Baseline up to 30 days post-treatment
  The relationship between tumor (or cell-free [cf]DNA) PIK3CA mutation status/loss of phosphatase and tensin homolog gene (PTEN) and response to treatment will be described using contingency tables. The concordance between cfDNA and PIK3CA mutation status will also be assessed using contingency tables at baseline and following study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States